CLINICAL TRIAL: NCT05787119
Title: Benefit of Augmented Reality Mirror Therapy in Addition to Conventional Management in Complex Regional Pain Syndrome of the Upper Extremity: a Single Case Experimental Design (SCED) Study.
Brief Title: Benefit of Augmented Reality Mirror Therapy in Addition to Conventional Management in Complex Regional Pain Syndrome of the Upper Extremity
Acronym: REFLEXION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NIMAO/2022-AD-01
Record Dates: First submitted 2023-03-10; First posted 2023-03-28 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Complex Regional Pain Syndromes
Keywords: Mirror Movement Therapy; Physical Therapy Modalities
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): 2 weeks Conventional therapy / 1 month ARMT / 4 weeks Conventional therapy
  Interventions: Other: Conventional therapy; Other: ARMT; Other: cortical reactivity; Other: Fluidity of movement
- Group 2 (Experimental): 3 weeks Conventional therapy / 1 month ARMT / 3 weeks Conventional therapy
  Interventions: Other: Conventional therapy; Other: ARMT; Other: cortical reactivity; Other: Fluidity of movement
- Group 3 (Experimental): 2.5 weeks Conventional therapy / 1 month ARMT / 3.5 weeks Conventional therapy
  Interventions: Other: Conventional therapy; Other: ARMT; Other: cortical reactivity; Other: Fluidity of movement

INTERVENTIONS:
Other: Conventional therapy — The CT consists of 1 session of 30 minutes of physical therapy (type of re-education established according to the pain at rest and during movement assessed every day) and 1 session of 30 minutes of occupational therapy (type of re-education established according to the pain at rest and during movement assessed every day). CT is performed 5 days a week.
Other: ARMT — The ARMT consists of 1 session of 30 minutes (type of rehabilitation established according to the pain at rest and during movement evaluated daily). ARMT is performed 5 days a week for 1 month.
Other: cortical reactivity — An electroencephalogram was taken at the start and end of the study to study cortical reactivity during the performance of 3 different tasks repeated 30 times: a resting task (consisting of looking at a cross on a screen), a motor imagery task (consisting of imagining performing wrist flexions/extensions) and a motor execution task (consisting of performing wrist flexions/extensions).
Other: Fluidity of movement — Motion capture at the start and end of the study to study the fluidity of movement during 3 different tasks repeated 30 times: a resting task (looking at a cross on a screen), a motor imagery task (imagining wrist flexions/extensions) and a motor execution task (performing wrist flexions/extensions).

SUMMARY:
Complex Regional Pain Syndrome (CRPS) is a "polymorphic joint and periarticular pain syndrome associated with various changes in sensitivity, vasomotor, sudomotor, muscular and trophic changes". The diagnostic criteria of the disease follow the Budapest criteria, namely (i) vasomotor disorders (temperature asymmetry, color changes), (ii) sudomotor/oedema (sweating changes, edema), (iii) sensory (hyperesthesia, allodynia, hyperalgesia) and (iv) motor/trophic (reduced joint mobility, weakness, tremor, dystonia, trophic disorders of skin, nails, hair).

Of the many treatments, augmented reality mirror therapy (ARMT), is novel in substituting a virtual environment for part of the real environment. This type of device has never been studied from a clinical point of view in the treatment of upper limb CRPS, whereas fMRI and clinical dissertation studies have suggested an improvement in neuroplasticity.

The aim of this study is to establish the clinical effects of ARMT on CRPS, and to evaluate its benefit within a conventional rehabilitation treatment (physiotherapy and occupational therapy).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient with CRPS of the upper limb according to the Budapest criteria.
* Patient newly treated at the Centre d'Evaluation et de Traitement de la Douleur of the CHU of Nîmes.
* Patient with a diagnosis of CRPS for more than 3 months

Exclusion Criteria:

* The subject is participating in a therapeutic study, or is in a period of exclusion determined by a previous study
* The subject unable to express consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient is pregnant, parturient or breastfeeding
* Patient with medically significant visual impairment that is incompatible with the practice of ARMT
* Patient with CRPS secondary to a stroke
* Patient with cognitive disorders (Montreal Cognitive Assessment scale less than 26)
* Patient with Unilateral Spatial Negligence according to the Bell's test
* Patient with arthrodesis of one of the joints of the upper limbs.
* Patient with an unhealed fracture of one of the upper limbs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in upper extremity motor function using ARMT versus CT alone | Every Monday and Thursday until study end (10 weeks)
  Change in Box and Block Test (BBT) score. The score will be compared between the right and left hand and against reference values according to age and sex.

SECONDARY OUTCOMES:
Improvement in clinical signs of CRPS using ARMT versus CT alone | Every Monday and Thursday until study end (10 weeks)
  Change in Complex regional pain syndrome Severity Score (CSS); score out of 16
Improvement in quality of life using ARMT versus CT alone | Every Monday and Thursday until study end (10 weeks)
  Change in EQ-5D-3L questionnaire score. The first part is a score out of 15 total (scoring out of 3 per item). The second part is a scale numbered 0 to 100 (0 being the worst health imaginable to 100 being the best health imaginable).
Improvement in global impression of change using ARMT versus CT alone | Every Monday and Thursday until study end (10 weeks)
  Change in Patient Global Impression of Change (PGIC) Questionnaire score. The measurement is between 1 and 7. It is a qualitative scale converted into a numerical scale.
Improvement in deep proprioceptive sensitivity of the upper limb using ARMT versus CT alone | Every Monday and Thursday until study end (10 weeks)
  Change in proprioceptive section of the Rivermead Assessment of Somatosensory Performance questionnaire score. 5 joints are tested 6 times. Thus for each joint, the score is out of 6, for a total score of 30.
Improvement of mental imagery ability using ARMT versus CT alone | Every Monday and Thursday until study end (10 weeks)
  Change in mental chronometry. Measured using a modified Box and Block Test to give a ratio = (real task time - imagined task time) / real task time
Improvement n perceived pain at movement and at rest using ARMT versus CT alone | Daily until study end (10 weeks)
  Change in pain, reported on a 0-10 visual analog scale
effectiveness of rehabilitation program adding TMRA device on cortical reactivity or Event related Potential (ERP) between pre- and post-treatment on pathological limb | Before Intervention (Day 0) and at the end of the study (10 weeks)
  Measurement of signal power amplitude (in microVolts) in motor imagery task and motor execution task compared with a resting task
evolution of cortical reactivity or event-related potential (ERP) between the healthy and pathological sides following a rehabilitation program adding a TMRA device. | at the end of the study (10 weeks)
  Amplitude of signal power (in microVolts) in motor imagery task and motor execution task compared with a resting task
effectiveness of a rehabilitation program adding a TMRA device on smoothness of movement on the pathological limb between pre- and post-treatment | Before Intervention (Day 0) and at the end of the study (10 weeks)
  Leap Motion Control motion capture device from Ultraleap Company (description)
To compare the smoothness of movement between the healthy and pathological side following a rehabilitation programme adding a TMRA device. | at the end of the study (10 weeks)
  Amplitude of signal power in motor imagery task and motor execution task compared with a resting task (descriptive, adimentional)
Correlate the power of cortical reactivity with fluidity of movement, function, mental chronometry, quality of life, global impression of change, proprioceptive sensitivity and clinical criteria of severity. | Before Intervention (Day 0) and at the end of the study (10 weeks)
  Correlation between 2 signals: cortical and motor for motor execution tasks (adimentional)
Correlate fluidity of movement with the power of cortical reactivity, function, mental chronometry, quality of life, global impression of change, proprioceptive sensitivity and clinical criteria of severity. | Before Intervention (Day 0) and at the end of the study (10 weeks)
  Multiple correlation (adimentional)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud DUPEYRON, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No